CLINICAL TRIAL: NCT03228043
Title: Apatinib With Postoperative Adjuvant Chemotherapy for Operable Colorectal Cancer
Brief Title: Apatinib for Resectable Colorectal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It's not possible to complete in our hospital.
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Principal Investigator, Yunhong Tian, Principal Investigator, Nanchong Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Apatinib in Colorectal Surgery
Record Dates: First submitted 2017-04-30; First posted 2017-07-24 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Apatinib; Outcome, Fatal; Colorectal Cancer; Surgery; Adjuvant Chemotherapy
Keywords: Apatinib; Outcome, Fatal; Colorectal Cancer; surgery; adjuvant chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib; Chemotherapy, Adjuvant

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib group (Experimental): Apatinib combined with CAPEOX program. Apatinib tablets: 500 mg po qd from the second cycle of chemotherapy. Oxaliplatin: Day 1, 130mg/m2, IV infusion. Capecitabine: Day 1-14, 1000mg/m2 Twice Daily, po. A total of 6 cycles, 3 weeks apart of chemotherapy.
  Interventions: Drug: Apatinib
- Control group (Placebo Comparator): CAPEOX program. Oxaliplatin: Day 1, 130mg/m2, IV infusion. Capecitabine: Day 1-14, 1000mg/m2 Twice Daily, po. A total of 6 cycles, 3 weeks apart of chemotherapy.
  Interventions: Drug: CAPEOX

INTERVENTIONS:
Drug: Apatinib — Apatinib combine with CAPEOX adjuvant chemotherapy for resectable colorectal
  Other Names: YN968D1
  Arms: Apatinib group
Drug: CAPEOX — CAPEOX adjuvant chemotherapy for resectable colorectal
  Other Names: adjuvant chemotherapy
  Arms: Control group

SUMMARY:
Objective: To compare the outcome of patients with colorectal cancer who treated with adjuvant therapy or Apatinib with adjuvant therapy postoperatively.

Language: English.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status score: 0-1.
2. All colorectal cancer patients underwent curative intent surgery
3. Patients in stage Ⅱ(Any T, N0, M0) with multiple high-risk factors or stage Ⅲ (any T, N1-2, M0) which confirmed by pathology.
4. Patients who did not receive other treatments for colorectal adenocarcinoma after surgery;
5. The main organ function is good, patients must meet the following requirements with 14 days before using Apatinib:

   * blood routine examination:

     * hemoglobin> 90 g / L (14 days without blood transfusion);
     * neutrophil count> 1.5 x 109 / L;
     * platelet count> 100 × 109 / L;
   * biochemical examination:

     * total bilirubin ≤ 1.5 × ULN (normal upper limit);
     * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2 × ULN;
     * Endogenous creatinine clearance ≥ 60 ml / min (Cockcroft-Gault formula);
   * Cardiac Doppler Ultrasonography: Left ventricular ejection fraction (LVEF) ≥ 50%.
6. The surgical incision has been healed, and no bleeding tendency;
7. Sign informed consent;
8. Compliance is good, family members agreed to accept survival follow-up.

Exclusion Criteria:

1. Patients with other malignancies, except for cured skin basal cell carcinoma and cervical cancer in situ.
2. Participated in other drug clinical trials within four weeks.
3. Have a variety of factors that affect oral medication (such as unable to swallow, chronic diarrhea and intestinal obstruction, etc.).
4. Have a history of bleeding, screening within 4 weeks before any serious grade to CTCAE4.0 3 degrees or more bleeding events.
5. Patients with central nervous system metastases or a history of central nervous system metastases before screening. For patients with suspected central nervous system metastases, CT or MRI examinations must be performed within 28 days prior to randomization to exclude central nervous system metastasis.
6. History of high blood pressure can not be controlled with a single antihypertensive drug therapy (With a systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg. A history of unstable angina within 3 months or a new diagnosis of angina within 6 months (Including QTcF: male ≥ 450 ms, female ≥470 ms) required long-term use of antiarrhythmic drugs and New York Heart Association classification ≥ Class II cardiac insufficiency.
7. Urinary protein ≥ ++ and urine protein> 1.0 g in 24 hours.
8. Patients with anastomotic fistula, pancreatic fistula or anastomotic stenosis and other serious postoperative complications.
9. Long-term non-healing wounds or bone fractures.
10. history of organ transplantation.
11. Imaging shows that the tumor has involved important vascular. Patients in high risk of fatal bleeding during treatment.
12. coagulation abnormalities, with bleeding tendency (14 days before randomization must meet: in the absence of anticoagulants, INR in normal range). application of anticoagulants or vitamin K antagonists such as warfarin, (1 mg orally, once daily) or low-dose aspirin (1 mg or less daily) at a prokaryotic time (INR) ≤ 1.5 Daily consumption of not more than 100 mg).
13. During the last year, the history of tachycardia / venous thrombosis events, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis (due to pre-chemotherapy intravenous thrombosis caused by intravenous thrombosis which have been cured ) And pulmonary embolism.
14. previous thyroid dysfunction, thyroid function can not be maintained within the normal range during medication.
15. with a history of psychiatric drug abuse and can not be prevented or have mental disorders.
16. Have a history of immunodeficiency, or suffer from other acquired, congenital immunodeficiency disease, or organ transplant history.
17. According to the researcher's judgment, there is a serious risk of compromising the patient's safety or affecting the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants recurrence-free survival | 1 year
  Number of Participants recurrence-free survival in intervention group and control group.
Number of Participants overall survival | 1 year
  Number of Participants overall survival in intervention group and control group.

SECONDARY OUTCOMES:
Number of Participants recurrence-free survival | 2 years
  Number of Participants recurrence-free survival in intervention group and control group.
Number of Participants overall survival | 2 years
  Number of Participants overall survival in intervention group and control group.

OTHER OUTCOMES:
Number of Participants recurrence-free survival | 3 years
  Number of Participants recurrence-free survival in intervention group and control group.
Number of Participants overall survival | 3 years
  Number of Participants overall survival in intervention group and control group.
Number of Participants recurrence-free survival | 4 years
  Number of Participants recurrence-free survival in intervention group and control group.
Number of Participants overall survival | 4 years
  Number of Participants overall survival in intervention group and control group.
Number of Participants recurrence-free survival | 5 years
  Number of Participants recurrence-free survival in intervention group and control group.
Number of Participants overall survival | 5 years
  Number of Participants overall survival in intervention group and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Yunhong Tian, Principal Investigator — Nanchong Central Hospital
Locations (1):
- Yunhong Tian, Nanchong, Sichuan, China

IPD SHARING:
Plan to Share IPD: No